CLINICAL TRIAL: NCT01492101
Title: The BEACON Study (Breast Cancer Outcomes With NKTR-102): A Phase 3 Open-Label, Randomized, Multicenter Study of NKTR-102 Versus Treatment of Physician's Choice (TPC) in Patients With Locally Recurrent or Metastatic Breast Cancer Previously Treated With an Anthracycline, a Taxane and Capecitabine
Brief Title: The BEACON Study (Breast Cancer Outcomes With NKTR-102)
Acronym: BEACON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-PIR-11
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Locally Recurrent Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NKTR-102 (Experimental)
  Interventions: Drug: NKTR-102
- Physician's Treatment of Choice (Active Comparator)
  Interventions: Drug: Treatment of Physician's Choice (TPC)

INTERVENTIONS:
Drug: NKTR-102 — 145 mg/m2 NKTR-102 will be delivered q21day as a 90-minute intravenous (IV) infusion on day 1 of each treatment cycle.
  Arms: NKTR-102
Drug: Treatment of Physician's Choice (TPC) — One of the following Treatment of Physician Choice will be administered per standard of care:
  eribulin, ixabepilone, vinorelbine, gemcitabine, paclitaxel, docetaxel, or nab-paclitaxel
  Arms: Physician's Treatment of Choice

SUMMARY:
The study is designed as an open-label, randomized, parallel, two arm, multicenter, international Phase 3 study in patients with recurrent or metastatic breast cancer previously treated with cytotoxic chemotherapy regimens.

The primary study objective is to compare overall survival of patients who receive NKTR-102 given once every 21 days to patients who receive treatment of Physician's Choice selected from a list of seven single-agent intravenous therapies.

ELIGIBILITY:
Inclusion Criteria (major highlights):

* Patient is an adult female with histologically or cytologically confirmed carcinoma of the breast for whom single-agent cytotoxic chemotherapy is indicated
* Patient can have either measurable or non-measurable disease by RECIST.
* Patient has received prior therapy (administered in the neoadjuvant, adjuvant and/or metastatic setting) with an anthracycline, a taxane and capecitabine
* Patient has minimum of 2 and a maximum of 5 prior cytotoxic chemotherapy regimens with the last dose administered within 6 months. A minimum of two chemotherapy regimens had to be for locally recurrent and/or metastatic disease. All therapy received prior to a diagnosis of metastatic disease (eg, neoadjuvant, adjuvant or repeated adjuvant therapy following a second resection) is counted as one regimen.
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematopoietic, liver and kidney functions.

Exclusion Criteria (major highlights):

* Patient with chemotherapy within 21 days, radiotherapy within 14 days, biological therapy with 14 days, hormonal therapy within 7 days and investigational therapy within 21 days prior to randomization.
* Patient with any major surgery within 28 days prior to randomization.
* Patient with concurrent use of biologic agents for the treatment of cancer including antibodies or any investigational agent(s).
* Patient with prior treatment for cancer with a camptothecin derivative.
* Patient with chronic or acute GI disorders resulting in diarrhea of any severity grade; patients who are using chronic anti-diarrheal supportive care to control diarrhea in the 28 days prior to randomization.
* Patient received pharmacotherapy for hepatitis B or C, tuberculosis or HIV.
* Patient with known cirrhosis diagnosed with Child-PUGH Class A or higher liver disease.
* Patient with prior malignancy (other than breast cancer) except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 5 years prior to randomization.
* Patient requiring daily use of oxygen supplementation in the 28 days prior to randomization.
* Patients with significant cardiovascular impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2011-12; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Hannah, MD, Study Director — Nektar Therapeutics
Locations (153):
- United States (88):
  - Arizona Oncology Associates, PC - NAHOA, Flagstaff, Arizona
  - Providence Health System - Southern California d/b/a Roy and Patricia Disney Family Cancer Center, Burbank, California
  - University of Southern California, Los Angeles, California
  - PMK Medical Group, Inc., DBA Ventura County Hematology Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Inc., Pasadena, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - University of California San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Kaiser Permanente, Vallejo, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Pre clinical Science Bldg LR3, Washington D.C., District of Columbia
  - Medstar, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Peachtree Hematology Oncology Consultants, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Summit Cancer Care, P.C., Savannah, Georgia
  - The University of Chicago Medicine, Chicago, Illinois
  - Oncology Specialists, Niles, Illinois
  - Illinois Cancer Care, P.C., Peoria, Illinois
  - IU Health Simon Cancer Center, Indianapolis, Indiana
  - Hall-Perrine Cancer Center, 3rd Floor, Cedar Rapids, Iowa
  - Kansas City Cancer Center, Overland Park, Kansas
  - Louisville Oncology Clinical Research Program, Louisville, Kentucky
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Frontier Cancer Center and Blood Institute, Billings, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hematology-Oncology Associates of Northern NJ, PA, Morristown, New Jersey
  - The cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cooper University Hospital, Voorhees Township, New Jersey
  - UNM Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Beth Israel Medical Center, New York, New York
  - Cornell University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Monte fiore, The Bronx, New York
  - Sciode Medical Associates, PLLC, d.b.a. Eastchester Center for Cancer Care, The Bronx, New York
  - Carolinas Hematology Oncology Associates, Charlotte, North Carolina
  - DUMC, Duke South, Durham, North Carolina
  - Sanford Research/USD, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Comprehensive Breast Cancer, Columbus, Ohio
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Cancer Centers of the Carolinas, Easley, South Carolina
  - Sanford Research/USD, Sioux Falls, South Dakota
  - The West Clinic, Memphis, Tennessee
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Abilene, Abilene, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology-Beaumont, Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology-Bedford, Bedford, Texas
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Texas Oncology-Fort Worth, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology-Lewisville, Lewisville, Texas
  - Texas Oncology-Mesquite, Mesquite, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology, P.A. - Plano, Plano, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Salem, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Cancer TEAM Bellin Health, Green Bay, Wisconsin
- Belgium (8):
  - Institut Jules Bordet, Brussels
  - GHdC - Site Notre Dame, Charleroi
  - Universtair Ziekenhuis Antwerpen, Edegem
  - UZ Gent Medische Oncologie, Ghent
  - UZ Leuven, Campus Gasthuisberg, trialbureau Algemene Medische Oncologie, Leuven
  - Centre Hospitalier Universitaire de Liège- Site du Sart Tilman, Liège
  - Centre Hospitalier Universitaire Ambroise Paré, Mons
  - GZA Ziekenhuizen, Campus St Augustinus, CLINICAL TRIALS ONCOLOGY, Wilrijk
- Canada (6):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Odette Cancer Centre OCC Clinical Research, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM-Hopital Notre-Dame, Montreal, Quebec
  - MUHC- Montreal General Hospital, Montreal, Quebec
  - Hôpital Charles-LeMoyne - CICM, Québec
- France (9):
  - Institut Bergonie Service Oncologie Médicale, Bordeaux
  - Sorecoh, Le Mans
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Service Pharmacie, Marseille
  - Centra Regional de Lutte contre le Cancer, Montpellier
  - Institut Curie, UGEC, Paris
  - Hopital Tenon Service oncologie médicale, Paris
  - Centre Régional de Lutte Contre le Cancer Nantes Atlantique René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Gustave Roussy, Villejuif
- Germany (7):
  - Klinikum St. Marien Amberg, Amberg
  - Onkoplus, Berlin
  - Oncoresearch, Dortmund
  - Universitaetsklinikum Erlangen, Erlangen
  - Wilhelm-Anton-Hospital gGmbH, Goch
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Ulm, Frauenklinik, Ulm
- Italy (5):
  - Istituto tumori Giovanni Paolo II-ospedale oncologico, Oncologia Medica e Sperimentale, Bari
  - Via Olgettina, Milan
  - Azienda Ospedaliero Universitaria Pisana, U.O. Oncologia Medica, Pisa
  - Oncologia Ospedale Infermi- Viale, Rimini
  - Istituto Nazionale tumori Regina Elena IRCCS, Roma
- Netherlands (3):
  - VUmc, Amsterdam
  - MUMC, Maastricht
  - Tweesteden Ziekenhuis, Tilburg
- Russia (5):
  - Leningrad Regional Oncology Dispensary, Kuz'molovskiy
  - State Institution "Russian Oncology Research Centre named after N.N. Blokhin RAMS", Moscow
  - Non-state Health Institution "Dorozhnaya Clinical Hospital of OAO "Russian Railways", Saint Petersburg
  - St. Petersburg State Budget Healthcare Institution "City Clinical Oncology Dispensary", Saint Petersburg
  - Scientific Research Oncology Institute named after N.N. Petrov, Saint Petersburg
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Samsung Medical Center, Irwon-dong, Seoul
  - Hematology-oncology Department, Ajou University Hospital, Sŏwŏn, Suwon
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Hematology-oncology Department, Ewha Womans University Mokdong Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital,, Soeul
- Spain (7):
  - Hospital Vall d'Hebron, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - MD Anderson Cancer Center Arturo, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Sant Joan de Reus, Tarragona
- United Kingdom (7):
  - Clinical Trials Unit, Velindre Cancer Centre, Cardiff
  - Beaston Oncology Center, Glasgow
  - St James University Hospital, Leeds
  - NCRN, London
  - The Christie Hospitals NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Cancer Clinical Trials Centre, Weston Park Hospital, Sheffield

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581
- [Derived] Cortes J, Rugo HS, Awada A, Twelves C, Perez EA, Im SA, Gomez-Pardo P, Schwartzberg LS, Dieras V, Yardley DA, Potter DA, Mailliez A, Moreno-Aspitia A, Ahn JS, Zhao C, Hoch U, Tagliaferri M, Hannah AL, O'Shaughnessy J. Prolonged survival in patients with breast cancer and a history of brain metastases: results of a preplanned subgroup analysis from the randomized phase III BEACON trial. Breast Cancer Res Treat. 2017 Sep;165(2):329-341. doi: 10.1007/s10549-017-4304-7. Epub 2017 Jun 13. PMID 28612225
- [Derived] Twelves C, Cortes J, O'Shaughnessy J, Awada A, Perez EA, Im SA, Gomez-Pardo P, Schwartzberg LS, Dieras V, Yardley DA, Potter DA, Mailliez A, Moreno-Aspitia A, Ahn JS, Zhao C, Hoch U, Tagliaferri M, Hannah AL, Rugo HS. Health-related quality of life in patients with locally recurrent or metastatic breast cancer treated with etirinotecan pegol versus treatment of physician's choice: Results from the randomised phase III BEACON trial. Eur J Cancer. 2017 May;76:205-215. doi: 10.1016/j.ejca.2017.02.011. Epub 2017 Mar 27. PMID 28360015
- [Derived] Perez EA, Awada A, O'Shaughnessy J, Rugo HS, Twelves C, Im SA, Gomez-Pardo P, Schwartzberg LS, Dieras V, Yardley DA, Potter DA, Mailliez A, Moreno-Aspitia A, Ahn JS, Zhao C, Hoch U, Tagliaferri M, Hannah AL, Cortes J. Etirinotecan pegol (NKTR-102) versus treatment of physician's choice in women with advanced breast cancer previously treated with an anthracycline, a taxane, and capecitabine (BEACON): a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2015 Nov;16(15):1556-1568. doi: 10.1016/S1470-2045(15)00332-0. Epub 2015 Oct 22. PMID 26482278

RESULTS

PARTICIPANT FLOW:
Groups:
- NKTR-102: NKTR-102: 145 mg/m2 NKTR-102 will be delivered q21day as a 90 minute intravenous (IV) infusion on day 1 of each treatment cycle.
- Physician's Treatment of Choice: Treatment of Physician's Choice (TPC): One of the following Treatment of Physician Choice will be administered per standard of care:
  eribulin ixabepilone vinorelbine gemcitabine paclitaxel docetaxel or nab-paclitaxel
Period: Overall Study
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Started | 429 | 423
Completed | 92 | 81
Not Completed | 337 | 342
Not completed — Death | 323 | 322
Not completed — Withdrawal by Subject | 14 | 18
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NKTR-102 | Physician's Treatment of Choice | Total
Number analyzed (Participants) | 429 | 423 | 852
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 341 | 342 | 683
  >=65 years | 88 | 81 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.29) | 55.2 (10.1) | 55.2 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 429 | 423 | 852
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 15 | 24
  South Korea | 43 | 42 | 85
  Netherlands | 1 | 1 | 2
  Belgium | 53 | 39 | 92
  United States | 198 | 180 | 378
  Italy | 10 | 12 | 22
  United Kingdom | 19 | 23 | 42
  France | 36 | 47 | 83
  Germany | 0 | 4 | 4
  Spain | 46 | 51 | 97
  Russia | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Overall Survival: Intention to Treat (ITT) Population
Description: Duration of OS was defined as the time from the date of randomisation to the date of death due to any cause. Subjects were followed until their date of death, loss to follow-up, withdrawal of consent for further follow-up for survival, or final database closure. OS was determined using the ITT population which included all subjects randomized into 1 of the 2 treatment arms. Subjects who were lost-to-follow-up or were not known to have died were censored at last date they were shown to be alive. Subjects who did not have any follow-up since the date of randomization were censored at the date of randomization.
Time Frame: 36 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 429 | 423
Months | 12.4 [11.0 to 13.6] | 10.3 [9.0 to 11.3]
Statistical Analysis 1: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Other — Two-sided log-rank test, stratified by geographic region, prior use of eribulin, and receptor status; p = 0.0835, Log Rank; Hazard Ratio, log = 0.872, 95% CI 2-sided [0.747 to 1.019]

2. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS): ITT Population
Description: PFS was defined as the time from the date of randomization to the earliest date of disease progression (assessed by the investigator according to RECIST version 1.1) or death due to any cause. PFS was determined using the ITT population which included all subjects randomized into 1 of the 2 treatment arms. For subjects whose disease did not progress or who did not die, the PFS time was censored at the time of the last tumor assessment that demonstrated lack of disease progression. For subjects who received new anti-cancer therapy, the PFS time was censored at the start of the new anti-cancer therapy.
Time Frame: Up to 38 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 429 | 423
Months | 2.4 [2.1 to 3.5] | 2.8 [2.1 to 3.5]
Statistical Analysis 1: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Superiority; p = 0.3017, Log Rank; Hazard Ratio (HR) = 0.926, 95% CI 2-sided [0.798 to 1.075]

3. Secondary Outcome: Clinical Benefit Rate (CBR): ITT Population
Description: CBR was defined as the proportion of subjects with a CR, PR, or stable disease (SD) for at least 6 months (≥ 182 days).
Time Frame: Up to 38 months.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 429 | 423
percentage of subjects | 20.5 [16.8 to 24.6] | 19.6 [15.9 to 23.7]

4. Secondary Outcome: Duration of Response (DOR): Efficacy Evaluable Population
Description: DOR was defined as the time from first documented CR or PR until the earliest evidence of disease progression or death from any cause. Subjects who were alive without documented disease progression per RECIST version 1.1 were censored at the date of last tumor assessment without disease progression or start of new anti-cancer therapy for the study disease.
Time Frame: Up to 38 months.
Population: The population analyzed for this outcome measure solely comprised of patients who achieved CR or PR per RECIST.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 58 | 61
Months | 3.9 [3.5 to 5.1] | 3.7 [2.1 to 3.9]

5. Secondary Outcome: Incidence of Dose Reductions: Safety Population
Description: Proportion of subjects who had a reduction in dose.
Time Frame: Up to 38 months.
Measure: Number; unit: percentage of subjects
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 425 | 406
percentage of subjects | 27.5 | 28.3

6. Secondary Outcome: Quality of Life Questionnaire-Core 30 (QLQ-C30) Individual Scale, Overall Score: ITT Population
Description: The QLQ-C30 is composed of 5 multi-item functional scales (physical, role, social, emotional and cognitive functioning), a global health status/QoL scale, 3 symptom scales (fatigue, nausea/vomiting, and pain), and 6 single items (financial impact, appetite loss, diarrhoea, constipation, insomnia and dyspnoea). Most items are scaled 1 to 4 (1 = not at all, 2 = a little, 3 = quite a bit, 4 = very much) except the items contributing to the global health status/QoL, which are 7-point questions (1 = very poor to 7 = excellent). Raw scores were transformed using a linear transformation to standardize the results so that scores range from 0 to 100. n=number of subjects who completed each individual scale. Note that for scores measuring function, a higher score represented a higher "better" level of functioning, while for scores measuring symptoms, a higher score represented a lower "worse" level of symptoms.
Time Frame: Up to 39 months
Population: 429 (ITT Population) 423 (ITT Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 429 | 423
units on a scale
  Global health status/QoL: number analyzed (Participants) | 421 | 405
  Global health status/QoL | 61.4 (21.76) | 58.0 (20.43)
  Physical functioning: number analyzed (Participants) | 422 | 406
  Physical functioning | 74.5 (19.72) | 72.3 (19.74)
  Role functioning: number analyzed (Participants) | 422 | 405
  Role functioning | 71.8 (26.81) | 67.3 (26.93)
  Emotional functioning: number analyzed (Participants) | 421 | 405
  Emotional functioning | 72.4 (21.86) | 71.9 (20.06)
  Cognitive functioning: number analyzed (Participants) | 421 | 405
  Cognitive functioning | 82.5 (18.7) | 81.2 (19.04)
  Social functioning: number analyzed (Participants) | 421 | 405
  Social functioning | 73.0 (26.69) | 71.0 (25.06)
  Fatigue: number analyzed (Participants) | 422 | 406
  Fatigue | 37.7 (23.68) | 41.3 (22.98)
  Nausea and vomiting: number analyzed (Participants) | 422 | 406
  Nausea and vomiting | 8.6 (13.39) | 9.9 (16.17)
  Pain: number analyzed (Participants) | 422 | 406
  Pain | 32.3 (27.2) | 35.3 (28.01)
  Dyspnoea: number analyzed (Participants) | 421 | 406
  Dyspnoea | 24.5 (27.44) | 23.6 (26.2)
  Insomnia: number analyzed (Participants) | 421 | 406
  Insomnia | 29.3 (28.94) | 31.5 (27.11)
  Appetite loss: number analyzed (Participants) | 422 | 406
  Appetite loss | 24.3 (27.55) | 26.6 (27.89)
  Constipation: number analyzed (Participants) | 422 | 403
  Constipation | 18.0 (25.9) | 21.0 (28.15)
  Diarrhoea: number analyzed (Participants) | 421 | 404
  Diarrhoea | 6.3 (13.64) | 5.6 (11.14)
  Financial difficulties: number analyzed (Participants) | 421 | 404
  Financial difficulties | 26.4 (31.29) | 21.9 (28.95)

7. Secondary Outcome: QLQ-C30 Individual Scale, Change Over Time: ITT Population
Description: The QLQ-C30 is composed of 5 multi-item functional scales (physical, role, social, emotional and cognitive functioning), a global health status/QoL scale, 3 symptom scales (fatigue, nausea/vomiting, and pain), and 6 single items (financial impact, appetite loss, diarrhea, constipation, insomnia and dyspnea). Most items are scaled 1 to 4 (1 = not at all, 2 = a little, 3 = quite a bit, 4 = very much) except the items contributing to the global health status/QoL, which are 7-point questions (from 1 = very poor to 7 = excellent). Raw scores were transformed using a linear transformation to standardize the results so that scores range from 0 to 100. n=number of subjects who completed each individual scale. Note that for scores measuring function, a higher score represented a higher "better" level of functioning, while for scores measuring symptoms, a higher score represented a lower "worse" level of symptoms.
Time Frame: From Baseline to Week 8, Week 16, Week 24, Week 32, Week 40, Week 48, Week 56.
Population: 429 (ITT Population) 423 (ITT Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 429 | 423
units on a scale
  Global health status/QoL: Week 8: number analyzed (Participants) | 337 | 311
  Global health status/QoL: Week 8 | -4.4 (22.57) | -4.7 (20.37)
  Global health status/QoL: Week 16: number analyzed (Participants) | 181 | 159
  Global health status/QoL: Week 16 | -2.5 (22.9) | -5.6 (21.86)
  Global health status/QoL: Week 24: number analyzed (Participants) | 116 | 90
  Global health status/QoL: Week 24 | -1.8 (24.99) | -6.6 (22.47)
  Global health status/QoL: Week 32: number analyzed (Participants) | 69 | 59
  Global health status/QoL: Week 32 | -0.2 (20.39) | -6.3 (26.66)
  Global health status/QoL: Week 40: number analyzed (Participants) | 48 | 31
  Global health status/QoL: Week 40 | -5.2 (22.27) | -2.6 (19.41)
  Global health status/QoL: Week 48: number analyzed (Participants) | 29 | 19
  Global health status/QoL: Week 48 | -2.3 (18.62) | -1.8 (20.71)
  Global health status/QoL: Week 56: number analyzed (Participants) | 26 | 15
  Global health status/QoL: Week 56 | 2.9 (17.79) | -11.1 (29.36)
  Physical functioning: Week 8: number analyzed (Participants) | 340 | 315
  Physical functioning: Week 8 | -4.9 (17.98) | -7.1 (17.4)
  Physical functioning: Week 16: number analyzed (Participants) | 181 | 159
  Physical functioning: Week 16 | -3.0 (20.63) | -7.0 (18.26)
  Physical functioning: Week 24: number analyzed (Participants) | 116 | 92
  Physical functioning: Week 24 | 0.3 (20.93) | -4.7 (15.9)
  Physical functioning: Week 32: number analyzed (Participants) | 68 | 60
  Physical functioning: Week 32 | -3.0 (18.88) | -8.5 (20.4)
  Physical functioning: Week 40: number analyzed (Participants) | 48 | 31
  Physical functioning: Week 40 | -1.9 (19.23) | -6.4 (18.81)
  Physical functioning: Week 48: number analyzed (Participants) | 30 | 19
  Physical functioning: Week 48 | 0.2 (17.66) | -7.4 (16.46)
  Physical functioning: Week 56: number analyzed (Participants) | 26 | 16
  Physical functioning: Week 56 | 2.2 (13.48) | -10.4 (24.27)
  Role functioning: Week 8: number analyzed (Participants) | 340 | 314
  Role functioning: Week 8 | -6.6 (27.26) | -8.3 (27.37)
  Role functioning: Week 16: number analyzed (Participants) | 180 | 159
  Role functioning: Week 16 | -4.8 (26.06) | -8.3 (24.41)
  Role functioning: Week 24: number analyzed (Participants) | 116 | 91
  Role functioning: Week 24 | -7.8 (33.3) | -10.8 (26.72)
  Role functioning: Week 32: number analyzed (Participants) | 68 | 60
  Role functioning: Week 32 | -9.7 (19.03) | -12.2 (29.81)
  Role functioning: Week 40: number analyzed (Participants) | 48 | 30
  Role functioning: Week 40 | -8.7 (30.94) | -7.8 (27.93)
  Role functioning: Week 48: number analyzed (Participants) | 30 | 19
  Role functioning: Week 48 | -3.1 (25.38) | -5.7 (21.7)
  Role functioning: Week 56: number analyzed (Participants) | 26 | 16
  Role functioning: Week 56 | -2.6 (17.12) | -9.4 (35.08)
  Emotional functioning: Week 8: number analyzed (Participants) | 338 | 313
  Emotional functioning: Week 8 | -0.5 (19.65) | -2.0 (19.95)
  Emotional functioning: Week 16: number analyzed (Participants) | 181 | 160
  Emotional functioning: Week 16 | 2.7 (18.93) | -1.6 (20.57)
  Emotional functioning: Week 24: number analyzed (Participants) | 116 | 91
  Emotional functioning: Week 24 | -0.6 (22.34) | -3.7 (18.95)
  Emotional functioning: Week 32: number analyzed (Participants) | 69 | 59
  Emotional functioning: Week 32 | -2.8 (21.02) | -7.6 (20.88)
  Emotional functioning: Week 40: number analyzed (Participants) | 48 | 31
  Emotional functioning: Week 40 | -1.4 (26.12) | 0.8 (19.11)
  Emotional functioning: Week 48: number analyzed (Participants) | 29 | 19
  Emotional functioning: Week 48 | 0.9 (21.37) | 1.2 (18.83)
  Emotional functioning: Week 56: number analyzed (Participants) | 26 | 15
  Emotional functioning: Week 56 | -3.6 (19.72) | -4.7 (25.29)
  Cognitive functioning: Week 8: number analyzed (Participants) | 339 | 313
  Cognitive functioning: Week 8 | -3.3 (18.46) | -3.2 (19.44)
  Cognitive functioning: Week 16: number analyzed (Participants) | 181 | 160
  Cognitive functioning: Week 16 | -1.4 (17.67) | -4.4 (20.81)
  Cognitive functioning: Week 24: number analyzed (Participants) | 116 | 91
  Cognitive functioning: Week 24 | -1.8 (17.26) | -2.2 (17.12)
  Cognitive functioning: Week 32: number analyzed (Participants) | 69 | 59
  Cognitive functioning: Week 32 | -4.6 (17.82) | -7.9 (20.14)
  Cognitive functioning: Week 40: number analyzed (Participants) | 48 | 31
  Cognitive functioning: Week 40 | -5.7 (18.61) | -3.5 (21.6)
  Cognitive functioning: Week 48: number analyzed (Participants) | 29 | 19
  Cognitive functioning: Week 48 | -4.6 (18.04) | 2.2 (17.75)
  Cognitive functioning: Week 56: number analyzed (Participants) | 26 | 15
  Cognitive functioning: Week 56 | -2.9 (18.25) | -6.7 (22.97)
  Social functioning: Week 8: number analyzed (Participants) | 339 | 313
  Social functioning: Week 8 | -4.9 (27.46) | -6.2 (24.04)
  Social functioning: Week 16: number analyzed (Participants) | 181 | 160
  Social functioning: Week 16 | 0.4 (27.57) | -6.4 (24.2)
  Social functioning: Week 24: number analyzed (Participants) | 116 | 90
  Social functioning: Week 24 | -3.4 (25.68) | -7.2 (24.1)
  Social functioning: Week 32: number analyzed (Participants) | 69 | 59
  Social functioning: Week 32 | -8.8 (20.61) | -7.2 (30.1)
  Social functioning: Week 40: number analyzed (Participants) | 48 | 31
  Social functioning: Week 40 | -9.7 (26.09) | -7.0 (20.98)
  Social functioning: Week 48: number analyzed (Participants) | 29 | 19
  Social functioning: Week 48 | -5.5 (17.86) | -6.6 (20.71)
  Social functioning: Week 56: number analyzed (Participants) | 26 | 15
  Social functioning: Week 56 | -3.2 (22.25) | -24.4 (29.96)
  Fatigue: Week 8: number analyzed (Participants) | 340 | 315
  Fatigue: Week 8 | 6.7 (22.88) | 6.6 (22.17)
  Fatigue: Week 16: number analyzed (Participants) | 180 | 161
  Fatigue: Week 16 | 3.7 (22.63) | 7.7 (22.84)
  Fatigue: Week 24: number analyzed (Participants) | 116 | 92
  Fatigue: Week 24 | 3.0 (26.51) | 3.6 (21.23)
  Fatigue: Week 32: number analyzed (Participants) | 69 | 60
  Fatigue: Week 32 | 5.0 (21.84) | 6.6 (24.25)
  Fatigue: Week 40: number analyzed (Participants) | 48 | 31
  Fatigue: Week 40 | 4.1 (26.65) | 2.3 (19.02)
  Fatigue: Week 48: number analyzed (Participants) | 30 | 19
  Fatigue: Week 48 | 0.9 (18.69) | 6.7 (14.53)
  Fatigue: Week 56: number analyzed (Participants) | 26 | 16
  Fatigue: Week 56 | 2.1 (19.57) | 4.5 (24.36)
  Nausea and vomiting: Week 8: number analyzed (Participants) | 340 | 315
  Nausea and vomiting: Week 8 | 12.8 (23.28) | 4.2 (21.94)
  Nausea and vomiting: Week 16: number analyzed (Participants) | 180 | 160
  Nausea and vomiting: Week 16 | 8.8 (19.85) | -2.0 (19.1)
  Nausea and vomiting: Week 24: number analyzed (Participants) | 116 | 92
  Nausea and vomiting: Week 24 | 7.2 (22.57) | -0.1 (16.55)
  Nausea and vomiting: Week 32: number analyzed (Participants) | 69 | 60
  Nausea and vomiting: Week 32 | 6.5 (14.21) | 3.5 (18.81)
  Nausea and vomiting: Week 40: number analyzed (Participants) | 48 | 31
  Nausea and vomiting: Week 40 | 4.5 (12.97) | 5.6 (23.61)
  Nausea and vomiting: Week 48: number analyzed (Participants) | 30 | 19
  Nausea and vomiting: Week 48 | 5.0 (13.77) | 3.9 (28.92)
  Nausea and vomiting: Week 56: number analyzed (Participants) | 26 | 16
  Nausea and vomiting: Week 56 | 8.0 (11.66) | 1.6 (23.02)
  Pain: Week 8: number analyzed (Participants) | 341 | 315
  Pain: Week 8 | -1.7 (26.08) | 2.4 (27.03)
  Pain: Week 16: number analyzed (Participants) | 182 | 161
  Pain: Week 16 | -5.0 (26.9) | 1.9 (27.8)
  Pain: Week 24: number analyzed (Participants) | 116 | 92
  Pain: Week 24 | -4.1 (29.35) | 2.1 (27.78)
  Pain: Week 32: number analyzed (Participants) | 69 | 60
  Pain: Week 32 | -1.0 (27.17) | 3.9 (32.49)
  Pain: Week 40: number analyzed (Participants) | 48 | 31
  Pain: Week 40 | 1.6 (31.82) | 1.3 (29.96)
  Pain: Week 48: number analyzed (Participants) | 30 | 19
  Pain: Week 48 | -0.8 (30.82) | -0.4 (25.23)
  Pain: Week 56: number analyzed (Participants) | 26 | 16
  Pain: Week 56 | -4.2 (22.88) | 0.5 (33.95)
  Dyspnoea: Week 8: number analyzed (Participants) | 339 | 313
  Dyspnoea: Week 8 | 0.7 (25.02) | 5.8 (24.59)
  Dyspnoea: Week 16: number analyzed (Participants) | 180 | 158
  Dyspnoea: Week 16 | -1.1 (26.34) | 4.6 (26.99)
  Dyspnoea: Week 24: number analyzed (Participants) | 116 | 92
  Dyspnoea: Week 24 | -2.0 (25.65) | 1.4 (20.47)
  Dyspnoea: Week 32: number analyzed (Participants) | 68 | 60
  Dyspnoea: Week 32 | 0 (24.77) | 8.6 (29.67)
  Dyspnoea: Week 40: number analyzed (Participants) | 48 | 30
  Dyspnoea: Week 40 | 2.4 (27.93) | 5.0 (25.95)
  Dyspnoea: Week 48: number analyzed (Participants) | 30 | 19
  Dyspnoea: Week 48 | -5.6 (26.38) | -0.9 (19.62)
  Dyspnoea: Week 56: number analyzed (Participants) | 26 | 14
  Dyspnoea: Week 56 | -7.1 (18.36) | -1.2 (22.13)
  Insomnia: Week 8: number analyzed (Participants) | 338 | 315
  Insomnia: Week 8 | -1.5 (28.1) | 3.3 (30.28)
  Insomnia: Week 16: number analyzed (Participants) | 180 | 160
  Insomnia: Week 16 | -1.4 (24.4) | 2.1 (27.2)
  Insomnia: Week 24: number analyzed (Participants) | 116 | 92
  Insomnia: Week 24 | -2.7 (31.77) | 1.3 (26.41)
  Insomnia: Week 32: number analyzed (Participants) | 68 | 59
  Insomnia: Week 32 | 1.5 (34.04) | 2.5 (30.14)
  Insomnia: Week 40: number analyzed (Participants) | 48 | 30
  Insomnia: Week 40 | 0 (31.51) | 4.4 (22.71)
  Insomnia: Week 48: number analyzed (Participants) | 30 | 19
  Insomnia: Week 48 | 2.8 (28.05) | 0.9 (34.01)
  Insomnia: Week 56: number analyzed (Participants) | 26 | 16
  Insomnia: Week 56 | -1.3 (35.57) | -1.0 (27.53)
  Appetite loss: Week 8: number analyzed (Participants) | 340 | 314
  Appetite loss: Week 8 | 11.6 (32.03) | 4.0 (30.26)
  Appetite loss: Week 16: number analyzed (Participants) | 180 | 159
  Appetite loss: Week 16 | 9.4 (32.16) | -2.1 (29.75)
  Appetite loss: Week 24: number analyzed (Participants) | 116 | 92
  Appetite loss: Week 24 | 4.6 (36.55) | -1.6 (30.57)
  Appetite loss: Week 32: number analyzed (Participants) | 69 | 60
  Appetite loss: Week 32 | 8.9 (35.42) | 0 (32.04)
  Appetite loss: Week 40: number analyzed (Participants) | 48 | 31
  Appetite loss: Week 40 | 6.9 (38.57) | 5.4 (38.58)
  Appetite loss: Week 48: number analyzed (Participants) | 30 | 18
  Appetite loss: Week 48 | 2.2 (34.67) | 13.0 (45.93)
  Appetite loss: Week 56: number analyzed (Participants) | 26 | 16
  Appetite loss: Week 56 | 14.7 (35.38) | 1.0 (39.19)
  Constipation: Week 8: number analyzed (Participants) | 337 | 310
  Constipation: Week 8 | 2.1 (29.95) | 6.7 (27.81)
  Constipation: Week 16: number analyzed (Participants) | 181 | 158
  Constipation: Week 16 | 0.2 (31.03) | 3.1 (30.96)
  Constipation: Week 24: number analyzed (Participants) | 116 | 90
  Constipation: Week 24 | 0.5 (29.65) | -2.0 (28.14)
  Constipation: Week 32: number analyzed (Participants) | 69 | 59
  Constipation: Week 32 | 4.6 (29.83) | 0.3 (26.53)
  Constipation: Week 40: number analyzed (Participants) | 48 | 31
  Constipation: Week 40 | 1.0 (28.44) | -3.2 (29.32)
  Constipation: Week 48: number analyzed (Participants) | 48 | 31
  Constipation: Week 48 | -0.6 (31.65) | 7.0 (33.48)
  Constipation: Week 56: number analyzed (Participants) | 26 | 15
  Constipation: Week 56 | 1.9 (34.42) | -4.4 (35.34)
  Diarrhoea: Week 8: number analyzed (Participants) | 339 | 311
  Diarrhoea: Week 8 | 10.2 (27.98) | 1.8 (16.87)
  Diarrhoea: Week 16: number analyzed (Participants) | 181 | 158
  Diarrhoea: Week 16 | 10.8 (26.97) | 3.4 (19.07)
  Diarrhoea: Week 24: number analyzed (Participants) | 114 | 89
  Diarrhoea: Week 24 | 9.4 (26.43) | 2.4 (16.39)
  Diarrhoea: Week 32: number analyzed (Participants) | 69 | 59
  Diarrhoea: Week 32 | 9.2 (21.3) | 0.8 (17.07)
  Diarrhoea: Week 40: number analyzed (Participants) | 48 | 30
  Diarrhoea: Week 40 | 8.3 (23.06) | 7.8 (27.93)
  Diarrhoea: Week 48: number analyzed (Participants) | 29 | 19
  Diarrhoea: Week 48 | 12.1 (22.23) | 0 (17.57)
  Diarrhoea: Week 56: number analyzed (Participants) | 26 | 15
  Diarrhoea: Week 56 | 4.5 (14.57) | 6.7 (31.37)
  Financial difficulties: Week 8: number analyzed (Participants) | 339 | 312
  Financial difficulties: Week 8 | -0.7 (22.87) | 0.6 (22.42)
  Financial difficulties: Week 16: number analyzed (Participants) | 181 | 159
  Financial difficulties: Week 16 | 0.8 (23.26) | 1.0 (22.48)
  Financial difficulties: Week 24: number analyzed (Participants) | 115 | 90
  Financial difficulties: Week 24 | 1.0 (21.09) | 4.6 (28.38)
  Financial difficulties: Week 32: number analyzed (Participants) | 69 | 59
  Financial difficulties: Week 32 | 1.2 (20.28) | 10.2 (26.81)
  Financial difficulties: Week 40: number analyzed (Participants) | 48 | 30
  Financial difficulties: Week 40 | 4.2 (21.61) | -1.7 (19.74)
  Financial difficulties: Week 48: number analyzed (Participants) | 29 | 19
  Financial difficulties: Week 48 | 0 (22.27) | 3.5 (18.9)
  Financial difficulties: Week 56: number analyzed (Participants) | 26 | 15
  Financial difficulties: Week 56 | -1.9 (21.25) | 5.6 (25.72)
Statistical Analysis 1: Comparison: NKTR-102 vs Physician's Treatment of Choice; Global health status/QoL: change from baseline to last assessment (Week 56); Test type: Equivalence — [2] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.635, F-test; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-2.65 to 4.33]
Statistical Analysis 2: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [3] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.1656, F-test; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-0.88 to 5.14]
Statistical Analysis 3: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [4] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.8356, F-test; Median Difference (Final Values) = 0.5, 95% CI 2-sided [-3.9 to 4.82]
Statistical Analysis 4: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [5] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.7727, F-test; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.88 to 3.88]
Statistical Analysis 5: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [6] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.7446, F-test; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.56 to 3.59]
Statistical Analysis 6: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [7] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.9169, F-test; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.0 to 4.45]
Statistical Analysis 7: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [8] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.9731, F-test; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-3.66 to 3.79]
Statistical Analysis 8: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [9] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p < 0.0001, F-test; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [3.88 to 10.67]
Statistical Analysis 9: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [10] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.1252, F-test; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-7.59 to 0.93]
Statistical Analysis 10: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [11] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.1717, F-test; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-6.83 to 1.22]
Statistical Analysis 11: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [12] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.5513, F-test; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.95 to 3.18]
Statistical Analysis 12: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [13] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.0009, F-test; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [3.57 to 13.72]
Statistical Analysis 13: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [14] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.2337, F-test; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-7.35 to 1.8]
Statistical Analysis 14: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [15] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p < 0.0001, F-test; Mean Difference (Final Values) = 10.3, 95% CI 2-sided [6.6 to 13.98]
Statistical Analysis 15: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [16] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.99, F-test; Mean Difference (Final Values) = 0, 95% CI 2-sided [-3.74 to 3.69]

8. Secondary Outcome: Quality of Life Questionnaire-breast Cancer-specific Module (BR23) Score Value: ITT Population
Description: The QLQ-BR23 incorporates 5 multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning, and 3 single items to assess sexual enjoyment, upset by hair loss and future perspective. Most items were scaled one to four except the items contributing to the global health status/QoL, which were seven-point questions. Raw scores were transformed using a linear transformation to standardize the results so that scores ranged from 0-100. Note that for scores measuring function, a higher score represented a higher "better" level of functioning, while for scores measuring symptoms, a higher score represented a lower "worse" level of symptoms.
Time Frame: Baseline
Population: 429 (ITT Population) 423 (ITT Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 429 | 423
units on a scale
  Body image: number analyzed (Participants) | 421 | 408
  Body image | 69.5 (28.94) | 69.9 (27.91)
  Sexual functioning: number analyzed (Participants) | 410 | 388
  Sexual functioning | 14.1 (19.24) | 13.3 (18.91)
  Sexual enjoyment: number analyzed (Participants) | 184 | 166
  Sexual enjoyment | 36.1 (29.25) | 34.2 (30.77)
  Future perspective: number analyzed (Participants) | 421 | 406
  Future perspective | 38.7 (30.53) | 36.1 (29.0)
  Systemic therapy side effects: number analyzed (Participants) | 423 | 408
  Systemic therapy side effects | 21.9 (16.37) | 22.3 (15.15)
  Breast symptoms: number analyzed (Participants) | 423 | 408
  Breast symptoms | 15.3 (21.55) | 15.8 (20.79)
  Arm symptoms: number analyzed (Participants) | 423 | 409
  Arm symptoms | 20.8 (23.4) | 22.2 (22.75)
  Upset by hair loss: number analyzed (Participants) | 244 | 225
  Upset by hair loss | 33.2 (34.15) | 30.5 (33.29)

9. Secondary Outcome: BR23 Score Change Over Time: ITT Population
Description: The QLQ-BR23 incorporates 5 multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning, and 3 single items assess sexual enjoyment, upset by hair loss and future perspective. Most items were scaled one to four except the items contributing to the global health status/QoL, which were seven-point questions. Raw scores were transformed using a linear transformation to standardize the results so that scores ranged from 0-100. Note that for scores measuring function, a higher score represented a higher "better" level of functioning, while for scores measuring symptoms, a higher score represented a lower "worse" level of symptoms.
Time Frame: Up to 38 months.
Population: 429 (ITT Population) 423 (ITT Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 429 | 423
units on a scale
  Body image: Week 8: number analyzed (Participants) | 342 | 310
  Body image: Week 8 | -0.8 (21.99) | -2.2 (20.49)
  Body image: Week 16: number analyzed (Participants) | 178 | 162
  Body image: Week 16 | -0.8 (24.31) | -2.3 (20.91)
  Body image: Week 24: number analyzed (Participants) | 113 | 96
  Body image: Week 24 | 0.8 (23.58) | -4.7 (20.97)
  Body image: Week 32: number analyzed (Participants) | 68 | 62
  Body image: Week 32 | -1.2 (26.27) | -0.3 (22.23)
  Body image: Week 40: number analyzed (Participants) | 48 | 30
  Body image: Week 40 | 3.3 (22.63) | -2.4 (20.98)
  Body image: Week 48: number analyzed (Participants) | 29 | 20
  Body image: Week 48 | -0.3 (25.47) | -1.1 (28.93)
  Body image: Week 56: number analyzed (Participants) | 27 | 16
  Body image: Week 56 | 3.9 (25.53) | -10.2 (26.61)
  Sexual functioning: Week 8: number analyzed (Participants) | 320 | 286
  Sexual functioning: Week 8 | -0.8 (16.07) | -2.2 (16.26)
  Sexual functioning: Week 16: number analyzed (Participants) | 166 | 143
  Sexual functioning: Week 16 | 0.1 (16.67) | -0.8 (17.28)
  Sexual functioning: Week 24: number analyzed (Participants) | 100 | 82
  Sexual functioning: Week 24 | -2.8 (16.72) | -1.4 (15.7)
  Sexual functioning: Week 32: number analyzed (Participants) | 61 | 57
  Sexual functioning: Week 32 | -2.2 (19.12) | -.7 (12.82)
  Sexual functioning: Week 40: number analyzed (Participants) | 43 | 25
  Sexual functioning: Week 40 | -5.4 (16.66) | 2.7 (16.27)
  Sexual functioning: Week 48: number analyzed (Participants) | 26 | 16
  Sexual functioning: Week 48 | -9.6 (19.68) | 1.6 (15.88)
  Sexual functioning: Week 56: number analyzed (Participants) | 25 | 15
  Sexual functioning: Week 56 | -5.3 (17.33) | 1.7 (13.06)
  Sexual enjoyment: Week 8: number analyzed (Participants) | 96 | 68
  Sexual enjoyment: Week 8 | 2.6 (19.84) | -4.2 (23.64)
  Sexual enjoyment: Week 16: number analyzed (Participants) | 51 | 33
  Sexual enjoyment: Week 16 | -0.3 (18.41) | -8.6 (21.7)
  Sexual enjoyment: Week 24: number analyzed (Participants) | 27 | 19
  Sexual enjoyment: Week 24 | 1.9 (29.72) | -3.5 (28.1)
  Sexual enjoyment: Week 32: number analyzed (Participants) | 17 | 13
  Sexual enjoyment: Week 32 | 2.0 (23.48) | -2.6 (20.24)
  Sexual enjoyment: Week 40: number analyzed (Participants) | 12 | 7
  Sexual enjoyment: Week 40 | -15.3 (29.69) | 7.1 (13.11)
  Sexual enjoyment: Week 48: number analyzed (Participants) | 6 | 5
  Sexual enjoyment: Week 48 | -27.8 (25.09) | 6.7 (14.91)
  Sexual enjoyment: Week 56: number analyzed (Participants) | 7 | 4
  Sexual enjoyment: Week 56 | -9.8 (16.27) | 0 (0)
  Future perspective: Week 8: number analyzed (Participants) | 342 | 309
  Future perspective: Week 8 | 3.5 (28.3) | 1.5 (27.21)
  Future perspective: Week 16: number analyzed (Participants) | 180 | 162
  Future perspective: Week 16 | 6.9 (27.17) | 3.6 (29.18)
  Future perspective: Week 24: number analyzed (Participants) | 113 | 94
  Future perspective: Week 24 | 9.3 (31.1) | 6.6 (29.55)
  Future perspective: Week 32: number analyzed (Participants) | 66 | 61
  Future perspective: Week 32 | 6.1 (30.19) | 4.4 (35.86)
  Future perspective: Week 40: number analyzed (Participants) | 49 | 30
  Future perspective: Week 40 | 7.1 (28.05) | 13.3 (37.75)
  Future perspective: Week 48: number analyzed (Participants) | 29 | 19
  Future perspective: Week 48 | 9.2 (27.31) | 6.1 (35.66)
  Future perspective: Week 56: number analyzed (Participants) | 25 | 16
  Future perspective: Week 56 | 16.0 (28.25) | -3.1 (45.22)
  Systemic therapy side effects: Week 8: number analyzed (Participants) | 345 | 312
  Systemic therapy side effects: Week 8 | 2.3 (13.74) | 7.9 (16.03)
  Systemic therapy side effects: Week 16: number analyzed (Participants) | 181 | 162
  Systemic therapy side effects: Week 16 | 3.0 (14.95) | 9.1 (17.7)
  Systemic therapy side effects: Week 24: number analyzed (Participants) | 115 | 96
  Systemic therapy side effects: Week 24 | 2.2 (15.55) | 6.9 (17.39)
  Systemic therapy side effects: Week 32: number analyzed (Participants) | 69 | 62
  Systemic therapy side effects: Week 32 | 3.5 (13.5) | 7.3 (18.01)
  Systemic therapy side effects: Week 40: number analyzed (Participants) | 49 | 30
  Systemic therapy side effects: Week 40 | 3.2 (16.62) | 10.1 (18.33)
  Systemic therapy side effects: Week 48: number analyzed (Participants) | 30 | 20
  Systemic therapy side effects: Week 48 | 0.3 (11.74) | 6.4 (15.68)
  Systemic therapy side effects: Week 56: number analyzed (Participants) | 27 | 16
  Systemic therapy side effects: Week 56 | -1.1 (11.06) | 6.8 (21.84)
  Breast symptoms: Week 8: number analyzed (Participants) | 342 | 310
  Breast symptoms: Week 8 | -1.7 (15.21) | -0.2 (13.82)
  Breast symptoms: Week 16: number analyzed (Participants) | 177 | 159
  Breast symptoms: Week 16 | -3.5 (14.6) | 0.1 (14.64)
  Breast symptoms: Week 24: number analyzed (Participants) | 115 | 97
  Breast symptoms: Week 24 | -4.8 (10.52) | -1.1 (13.48)
  Breast symptoms: Week 32: number analyzed (Participants) | 69 | 60
  Breast symptoms: Week 32 | -2.5 (14.26) | -2.8 (13.63)
  Breast symptoms: Week 40: number analyzed (Participants) | 48 | 30
  Breast symptoms: Week 40 | -1.9 (14.59) | -0.2 (11.02)
  Breast symptoms: Week 48: number analyzed (Participants) | 29 | 20
  Breast symptoms: Week 48 | -2.7 (12.16) | 0 (13.79)
  Breast symptoms: Week 56: number analyzed (Participants) | 26 | 16
  Breast symptoms: Week 56 | -3.4 (13.28) | 2.5 (12.15)
  Arm symptoms: Week 8: number analyzed (Participants) | 342 | 312
  Arm symptoms: Week 8 | -3.0 (16.72) | -0.9 (15.01)
  Arm symptoms: Week 16: number analyzed (Participants) | 178 | 159
  Arm symptoms: Week 16 | -5.1 (17.24) | 1.1 (18.24)
  Arm symptoms: Week 24: number analyzed (Participants) | 115 | 97
  Arm symptoms: Week 24 | -4.9 (20.06) | -0.3 (19.56)
  Arm symptoms: Week 32: number analyzed (Participants) | 69 | 60
  Arm symptoms: Week 32 | -4.4 (18.39) | -0.5 (19.03)
  Arm symptoms: Week 40: number analyzed (Participants) | 48 | 30
  Arm symptoms: Week 40 | -6.0 (21.86) | 5.2 (18.39)
  Arm symptoms: Week 48: number analyzed (Participants) | 29 | 20
  Arm symptoms: Week 48 | -5.6 (20.89) | -1.4 (12.98)
  Arm symptoms: Week 56: number analyzed (Participants) | 26 | 16
  Arm symptoms: Week 56 | -5.6 (19.44) | -1.4 (12.98)
  Upset by hair loss: Week 8: number analyzed (Participants) | 102 | 122
  Upset by hair loss: Week 8 | -4.7 (32.28) | 0.1 (28.63)
  Upset by hair loss: Week 16: number analyzed (Participants) | 54 | 58
  Upset by hair loss: Week 16 | 8.3 (33.61) | 2.9 (31.24)
  Upset by hair loss: Week 24: number analyzed (Participants) | 37 | 38
  Upset by hair loss: Week 24 | 6.8 (35.02) | 3.5 (30.3)
  Upset by hair loss: Week 32: number analyzed (Participants) | 17 | 22
  Upset by hair loss: Week 32 | 6.9 (31.76) | -2.3 (29.68)
  Upset by hair loss: Week 40: number analyzed (Participants) | 20 | 14
  Upset by hair loss: Week 40 | -4.2 (30.05) | 20.2 (29.37)
  Upset by hair loss: Week 48: number analyzed (Participants) | 7 | 10
  Upset by hair loss: Week 48 | -16.7 (31.91) | 21.7 (36.89)
  Upset by hair loss: Week 56: number analyzed (Participants) | 8 | 5
  Upset by hair loss: Week 56 | -14.6 (30.13) | 16.7 (44.1)
Statistical Analysis 1: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [17] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.5833, F-test; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.42 to 4.29]
Statistical Analysis 2: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [18] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.3098, F-test; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-1.24 to 3.9]
Statistical Analysis 3: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [19] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.6264, F-test; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-3.39 to 5.63]
Statistical Analysis 4: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [20] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.0003, F-test; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-7.11 to -2.1]
Statistical Analysis 5: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [21] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.2473, F-test; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-3.84 to 0.99]
Statistical Analysis 6: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [22] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.0333, F-test; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-5.54 to -0.23]
Statistical Analysis 7: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [23] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.2575, F-test; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-12.2 to 3.28]
Statistical Analysis 8: Comparison: NKTR-102 vs Physician's Treatment of Choice; Test type: Equivalence — [24] - Analysis of variance with change from baseline in linear transformed score at the last visit as the dependent variable and treatment arm, geographic region, prior use of eribulin, and receptor status as fixed effects; p = 0.1072, F-test; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [-1.22 to 12.34]

10. Secondary Outcome: Population Mean ± Standard Deviation (SD) Area Under the Concentration-Time Curve (AUC) for NKTR-102 and Metabolites After Multiple Administration of 145 mg/m^2 NKTR-102 [25]
Description: Plasma concentrations of NKTR-102 and its major metabolites irinotecan, SN38, SN38G, and APC were measured using validated analytical methods. The population pharmacokinetic (PK) model-derived mean AUC values were computed by integration from t = 0 (start of first dose) to 21 days after the last dose. Integration was implemented using a separate compartment defined as the amount of drug or metabolite in the central compartment divided by the model-estimated volume of distribution.
Time Frame: Up to 38 months.
Measure: Mean (Standard Deviation); unit: μg·h/mL
Arm/Group | NKTR-102
Number analyzed (Participants) | 95
μg·h/mL
  NKTR-102 | 4619 (4874)
  Irinotecan | 18.8 (22.1)
  SN38 | 5.32 (6.74)
  SN38G | 40.6 (39.2)
  APC | 4.0 (5.1)

11. Secondary Outcome: Population Mean ± SD Maximum Plasma Concentration (Cmax) for NKTR-102 and Metabolites After Multiple Administration of 145 mg/m^2 NKTR-102 [26]
Description: Plasma concentrations of NKTR-102 and its major metabolites irinotecan, SN38, SN38G, and APC were measured using validated analytical methods. The population PK model-derived mean Cmax values were computed by integration from t = 0 (start of first dose) to 21 days after the last dose. Integration was implemented using a separate compartment defined as the amount of drug or metabolite in the central compartment divided by the model-estimated volume of distribution.
Time Frame: Up to 38 months.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NKTR-102
Number analyzed (Participants) | 95
ng/mL
  NKTR-102 | 62701 (14576)
  Irinotecan | 138 (61.8)
  SN38 | 4.45 (1.82)
  SN38G | 47.7 (43.1)
  APC | 7.3 (6.7)

12. Secondary Outcome: Population Mean ± SD Elimination Half-life (t½) for NKTR-102 After Multiple Administration of 145 mg/m^2 NKTR-102 [27]
Description: Plasma concentrations of NKTR-102 and its major metabolites irinotecan, SN38, SN38G, and APC were measured using validated analytical methods. The population PK model-derived mean t½ values were computed by integration from t = 0 (start of first dose) to 21 days after the last dose. Integration was implemented using a separate compartment defined as the amount of drug or metabolite in the central compartment divided by the model-estimated volume of distribution. The t½ of all analytes was primarily driven by NKTR-102. Thus, the NKTR-102 t½ of 37 days also applies to all NKTR-102 metabolites.
Time Frame: Up to 38 months.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NKTR-102
Number analyzed (Participants) | 95
days | 36.8 (1.4)

13. Secondary Outcome: Objective Response Rate (ORR): Efficacy Evaluable Population
Description: ORR was defined as the proportion of subjects with a complete response (CR) or a partial response (PR), assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 The analyses were performed for subjects in the efficacy evaluable population who had measurable disease as determined by the investigator at baseline.
Time Frame: Up to 38 months.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NKTR-102 | Physician's Treatment of Choice
Number analyzed (Participants) | 354 | 358
percentage of subjects | 16.4 [12.7 to 20.7] | 17.0 [13.3 to 21.3]

ADVERSE EVENTS:
Time Frame: Up to 38 months.
Description: Safety Population NKTR-102 = 425; TPC = 406
Arm/Group | NKTR-102 | Physician's Treatment of Choice
All-Cause Mortality (participants affected / at risk) | 323/425 | 322/406
Serious Adverse Events (participants affected / at risk) | 128/425 | 129/406
Other Adverse Events (participants affected / at risk) | 417/425 | 404/406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-102 (N=425) | Physician's Treatment of Choice (N=406)
Aortic stenosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 10
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pyrexia (General disorders) | 3 | 5
General physical health deterioration (General disorders) | 3 | 3
Asthenia (General disorders) | 1 | 3
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 1
Generalised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Clostridium test positive (Investigations) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 6
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Brain oedema (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 1
Hepatic encephalopathy (Nervous system disorders) | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cholinergic syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgraphia (Nervous system disorders) | 1 | 0
Gliosis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Spinal chord compression (Nervous system disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 2
Vomiting (Gastrointestinal disorders) | 10 | 6
Ascites (Gastrointestinal disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 3 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 4 | 3
Bronchitis (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 1 | 3
Device related infection (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 2
Escherichia sepsis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 1 | 1
Abscess intestinal (Infections and infestations) | 1 | 0
Acute haemorrhagic conjunctivitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Breast infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Moraxella infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-102 (N=425) | Physician's Treatment of Choice (N=406)
Weight decreased (Investigations) | 57 (65) | 24 (25)
Neutrophil count decreased (Investigations) | 26 (41) | 50 (126)
Aspartate aminotransferase increased (Investigations) | 23 (24) | 29 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 58 (68) | 70 (87)
Cough (Respiratory, thoracic and mediastinal disorders) | 59 (64) | 52 (55)
Neutropenia (Blood and lymphatic system disorders) | 92 (174) | 126 (244)
Anaemia (Blood and lymphatic system disorders) | 64 (83) | 82 (105)
Dizziness (Nervous system disorders) | 55 (75) | 41 (51)
Dysgeusia (Nervous system disorders) | 34 (41) | 28 (44)
Neuropathy peripheral (Nervous system disorders) | 9 (9) | 50 (62)
Vision blurred (Eye disorders) | 68 (161) | 12 (13)
Fatigue (General disorders) | 145 (241) | 130 (163)
Asthenia (General disorders) | 91 (142) | 114 (170)
Pyrexia (General disorders) | 30 (39) | 63 (98)
Oedema peripheral (General disorders) | 20 (22) | 42 (49)
Insomnia (Psychiatric disorders) | 29 (45) | 33 (35)
Anxiety (Psychiatric disorders) | 20 (26) | 22 (23)
Nausea (Gastrointestinal disorders) | 255 (478) | 155 (249)
Diarrhoea (Gastrointestinal disorders) | 277 (1202) | 79 (128)
Vomiting (Gastrointestinal disorders) | 172 (342) | 72 (109)
Constipation (Gastrointestinal disorders) | 112 (167) | 126 (152)
Abdominal pain (Gastrointestinal disorders) | 89 (147) | 47 (52)
Abdominal pain upper (Gastrointestinal disorders) | 56 (71) | 37 (45)
Dyspepsia (Gastrointestinal disorders) | 34 (45) | 32 (50)
Stomatitis (Gastrointestinal disorders) | 17 (23) | 34 (43)
Alopecia (Skin and subcutaneous tissue disorders) | 44 (49) | 95 (102)
Rash (Skin and subcutaneous tissue disorders) | 23 (28) | 24 (28)
Myalgia (Musculoskeletal and connective tissue disorders) | 26 (30) | 59 (89)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (45) | 39 (41)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (35) | 42 (55)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (32) | 35 (43)
Bone pain (Musculoskeletal and connective tissue disorders) | 17 (20) | 35 (38)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 25 (28) | 26 (29)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 (28) | 26 (29)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 26 (31)
Decreased appetite (Metabolism and nutrition disorders) | 130 (169) | 98 (116)
Hypokalaemia (Metabolism and nutrition disorders) | 39 (54) | 37 (39)
Dehydration (Metabolism and nutrition disorders) | 34 (39) | 19 (25)
Urinary tract infection (Infections and infestations) | 26 (27) | 26 (28)
Upper respiratory tract infection (Infections and infestations) | 15 (18) | 27 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.